CLINICAL TRIAL: NCT06887725
Title: The Effect of Exercise Training on Knee Joint Proprioception in Patients With Rheumatoid A Exercise Training on Knee Joint Proprioception in Patients With Rheumatoid Arthritisrthritis
Brief Title: Exercise Training and Knee Joint Proprioception in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysima Barlak (Other)
Collaborators: Hacettepe University (Other); Hasan Kalyoncu University (Other)
Responsible Party: Sponsor-Investigator, Aysima Barlak, PT, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/140
Record Dates: First submitted 2025-03-16; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2022-12

CONDITIONS: Rheumatic Arthritis
Keywords: exercise; proprioception; biopsychosocial model; knee; muscle strength
MeSH Terms: conditions — Rheumatic Fever; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Group (Experimental)
  Interventions: Other: Exercise
- Kontrol Group (No Intervention)

INTERVENTIONS:
Other: Exercise — The Cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı-BETY) is an innovative exercise approach developed based on the biopsychosocial model. The parameters that form the basis of BETY are function-oriented core stabilization exercises, information management in pain, information management in mood, and information management in sexuality. BETY was shaped by the feedback of individuals with rheumatism who participated in regular exercise sessions for years and was introduced to the literature as a treatment method aiming to create changes in the cognitive structures of patients through exercise.
  Arms: Training Group

SUMMARY:
Rheumatoid arthritis (RA) is a chronic disorder that affects 0.5% to 1% of adults and is the result of an autoimmune attack against joint tissues. In recent years, advances in anti-rheumatoid drugs and treatment strategies have improved the health status of patients with RA. However, many patients do not achieve disease remission and experience progressive functional impairment. According to 2003 data from the National Health Interview Survey in the United States, by 2030, approximately 25% of adults aged 18 years and older are expected to have doctor-diagnosed arthritis, and 9.3% of adults are expected to have arthritis-related activity limitations.

In order for patients with RA to perform activities of daily living, it is very important for them to maintain their balance, i.e., their sense of proprioception. It is known that knee proprioception is decreased in RA. In addition, the presence of pain, decreased muscle strength, and functionality in patients with RA lead many of them to adopt a sedentary lifestyle.

The main aim of this study was to evaluate the effects of exercise training on knee joint proprioception in individuals with RA. In addition, it also aims to examine how exercise training improves pain, functionality, performance, fear of falling, biopsychosocial status, and quality of life. The importance of this research is that it provides more scientific data for improving knee joint proprioception in individuals with RA and guides clinical practice. It is also expected to contribute to the development of a comprehensive approach to improving the quality of life of patients by demonstrating not only the physical but also the psychological and functional effects of exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with RA
* Being able to walk
* Being between the ages of 40-65.
* Accepting to participate in the study and approving the informed consent form.
* Being literate and able to use technological devices.

Exclusion Criteria:

* Having acute inflammatory pathology in the knee joint.
* Knee arthroplasty surgery.
* Intra-articular or systemic corticosteroid use in the last 3 months.
* Having participated in an FTR program in the last 3 months.
* Advanced musculoskeletal, cardiac or peripheral vascular disease.
* Significant system or organ failure.
* Having a disease that will affect cognitive functions such as Alzheimer's disease or dementia

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Cognitive Exercise Therapy Approach (BETY)- Biopsychosocial Questionnaire | 3 mounths
  it is a 30-item Likert-type scale developed through repeated statistics of feedback from rheumatic individuals who have participated in exercise sessions for many years, expressing the healing characteristics. It evaluates the individual from a biopsychosocial perspective with the subheadings of pain, functionality-fatigue, mood, sociability, sexuality and sleep. It is scored between 0 and 120. BETY-BQ evaluates the individual from a holistic perspective with six subheadings: pain (5 items), functionality (9 items), mood (10 items), sociability (3 items), sexuality (2 items) and sleep (1 item). A high score indicates a low biopsychosocial status.

SECONDARY OUTCOMES:
Proprioception of the knee joint | 3 mounths
  Joint position sense was evaluated for proprioception measurement. All measurements were performed by a sports physician using a Biodex System III Isokinetic Dynamometer (Biodex Corp, Shirley, NY). For the reproduction test, which evaluates joint position sense, the passive method in the sitting position was used. The evaluation was performed for 30° and 60° knee flexion angles.
Health Assessment Questionnaire (HAQ) | 3 mounths
  It is a scale developed to question functional inadequacy in daily living activities. The scale questions a total of 8 activities, including dressing, sitting up, eating, walking, hygiene, reaching out, grasping and daily tasks, and consists of 20 questions. Each question is scored between 0 and 3. High scores indicate a decrease in the individual's functionality.
Hospital Anxiety Depression Scale (HADS) | 3 mounths
  It is a scale consisting of 14 questions (7 questions about depression, 7 questions about anxiety) that the individual is asked to answer by thinking about the last few days, and is scored between 0 and 3. The cut-off values of the scale are 10 for the anxiety subscale and 7 for the depression subscale. High total scores indicate high levels of anxiety or depression
WOMAC Osteoarthritis Index | 3 mounths
  WOMAC assesses pain, endurance and physical functioning, functional status and stiffness. This scale has gained increasing acceptance in the assessment of OA since its introduction in 1986. The pain subscale includes five items asking about pain with activity, at rest and at night. The stiffness heading includes two questions. The functional status heading includes an assessment of difficulty in 17 different activities. The items are scored from 0 to 4 according to difficulty and the degree of pain and stiffness felt, with a higher total score indicating greater severity of the disease.
McGill pain scale short form (SF McGill) | 3 mounths
  The form consists of three parts. In the first part, 11 of the 15 descriptive word groups evaluate the sensory and 4 evaluate the perceptual dimension of pain. These descriptive words are rated on an intensity scale from 0 to 3 (0=None, 1=Mild, 2=Moderate, 3=Very). In the first part of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score and total pain score. The second part of the form includes five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. In the third part, the patient's current pain intensity is assessed using a visual analogy scale (VAS).
Time Up and Go Test | 3 mounths
  It is a test that evaluates fall risk and mobility in the elderly. With this test, the time (sec.) for individuals to get up from a chair, walk a distance of 3 meters and sit back on the chair was measured. A trial test was performed once. Then the test was performed twice and the average of the two measurements was taken.
10-step stair climbing test | 3 mounths
  10-step stair climbing test:It is a test that evaluates the individual's stair climbing activity, lower extremity strength and dynamic balance.
  On a staircase with a railing, the 9th step is marked and the individual is asked to climb up and down as fast as he/she can and this time (sec) is measured with a stopwatch.
6 min walk test | 3 mounths
  This is a submaximal exercise test used to determine exercise capacity.
Fall efficacy scale | 3 mounths
  Developed in 1990 by Tinetti et al., it assesses a person's perception of stability and fear of falling during daily activities indoors. It consists of 10 items, answers are scored between 1 and 10. A score above 70 indicates fear of falling
World health organization quality of life scale-short form (WHOQOL-BREF) | 3 mounths
  Developed by the World Health Organization (WHO), the scale has two versions: long (WHOQOL-100) and short (WHOQOL-BREF). The WHOQOL-BREF scale consists of a total of 26 questions, 24 of which question perceived quality of life and 2 of which question perceived health status. It consists of 4 domains: physical, psychological, social relations and environmental domains. Since each domain independently expresses the quality of life in its own domain, domain scores are calculated between 4 and 20. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akgoz A, Yakut Y, Tufekci O, Aktas BE, Sari EO, Barlak A, Bayramlar K, Apras Bilgen S, Korkusuz F, Unal E. Biopsychosocial model-based exercise improves muscle strength, proprioception, pain, function, and quality of life in rheumatoid arthritis patients with knee involvement: a randomized controlled clinical tiral. Rheumatol Int. 2025 Sep 6;45(9):221. doi: 10.1007/s00296-025-05976-3. No abstract available. PMID 40913677